CLINICAL TRIAL: NCT04410939
Title: COVID-19 PCR Test Results in Asymptomatic Pregnants Admitted for Birth and Other Interventions in Our Clinic
Brief Title: COVID-19 PCR Test Results in Asymptomatic Pregnants
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Gpolat1
Record Dates: First submitted 2020-05-22; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Asymptomatic Pregnant
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Reverse transcription polymerase chain reaction — PCR test is performed from the oropharyngeal and nasal swab samples taken before admission to each pregnant to prevent contamination from the pregnant women hospitalized in this clinic. In addition, the same test is done before each operation and before the operation. The aim of the study is to scan these tests retrospectively and to determine the rate of positive COVID-19 cases in asymptomatic pregnant women. The results will determine the importance of the measures to be taken in the pregnant and undergoing pregnant women.

SUMMARY:
In order to prevent contamination from the pregnant women hospitalized in this clinic, the RT-PCR test is performed from the oropharyngeal and nasal swab sample taken before hospitalization. In addition, the same test is done before each operation and before the operation. The aim of the study is to scan these tests retrospectively and to determine the rate of positive COVID-19 cases in asymptomatic pregnant women. The results will determine the importance of the measures to be taken in the pregnant women who undergo intervention.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic pregnant women who will give birth in this clinic, dilatation and curettage due to missed abortion, cerclage due to cervical insufficiency, medical evacuation due to fetal anomaly, and routine PCR test taken for service for some treatments.

Exclusion Criteria:

* Having any COVID-19 infection symptoms (fever, cough, weakness, shortness of breath, sore throat, etc.)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients who apply to Istanbul Medipol University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Rate of positive COVID-19 cases in asymptomatic pregnant women | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Sutton D, Fuchs K, D'Alton M, Goffman D. Universal Screening for SARS-CoV-2 in Women Admitted for Delivery. N Engl J Med. 2020 May 28;382(22):2163-2164. doi: 10.1056/NEJMc2009316. Epub 2020 Apr 13. No abstract available. PMID 32283004